CLINICAL TRIAL: NCT06640855
Title: Academic Education of Midwifes in Germany - Teaching in the Field of Maternal and Infant Oral Health
Status: Completed | Type: Observational
Sponsor: Jana Biermann (Other)
Responsible Party: Sponsor-Investigator, Jana Biermann, Dr. med. dent., University Medical Center Goettingen
Organization: University Medical Center Goettingen (Other)
Other Study IDs: 24/8/24
Record Dates: First submitted 2024-09-25; First posted 2024-10-15 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Education, Medical
Keywords: dental education, midwife, midwifery

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this study is to learn about teaching of maternal and infant oral health in the recently implemented degree program Midwifery B.Sc. in Germany. The main questions it aims to answer are:

What contents regarding maternal and infant oral health are taught? How is teaching in the field of maternal and infant oral health organized? Study coordinators of all study locations of Midwifery B.Sc. in Germany are asked to participate in an online survey once.

ELIGIBILITY:
Inclusion Criteria:

* Returned questionnaire

Exclusion Criteria:

* Questionnaire not returned

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study coordinators of all academic locations for Midwifery B.Sc. in Germany
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Online-Questionnaire | 10 minutes
  Completion of a web based questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Preventive Dentistry, Periodontology and Cariology University Medical Center Goettingen, Göttingen, Germany